CLINICAL TRIAL: NCT01510366
Title: The Phase Ⅲ Clinical Trial Protocol for the Inactivated Poliomyelitis Vaccine Made From Sabin Strains
Brief Title: The Clinical Trial Protocol for the Inactivated Poliomyelitis Vaccine Made From Sabin Strains(Sabin IPV)
Acronym: IPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government); National Institute for the Control of Pharmaceutical and Biological Products, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMBCAMS-03; 2011L01484 (Other: China state food and drug adminstration)
Record Dates: First submitted 2012-01-06; First posted 2012-01-16 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Poliomyelitis
Keywords: Inactivated Poliomyelitis Vaccine; Sabin Strains; poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Inactivated Poliomyelitis Vaccine (Sabin strains) 3 x 0.5ml intramuscular injections.
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strains)
- Cohort 2: (Experimental): Inactivated Poliomyelitis Vaccine (Salk strains) 3 x 0.5ml intramuscular injections.
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Salk strains)

INTERVENTIONS:
Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) — Inactivated Poliomyelitis Vaccine (Sabin strains) 3 x 0.5ml intramuscular injections, one month apart.
  Other Names: Sabin IPV
  Arms: Cohort 1
Biological: Inactivated Poliomyelitis Vaccine (Salk strains) — Inactivated Poliomyelitis Vaccine (Salk strains)3 x 0.5ml intramuscular injections, one month apart.
  Other Names: Salk IPV or cIPV
  Arms: Cohort 2:

SUMMARY:
Based on pre-clinical trial and phase 1 and phase 2 clinical data and principle of GCP, the objective of phase Ⅲ clinical trial is to evaluate safety and immunogenicity of Inactivated Poliomyelitis Vaccine made from Sabin Strains(Sabin IPV).

DETAILED DESCRIPTION:
The Sabin IPV was manufactured with poliovirus type 1, 2, 3 Sabin strains and Vero cells by microcarrier culture in 550 liter bioreactors. The virus suspension was harvested, ultra-concentrated, purified and inactivated with formalin. The D Ag contents of Sabin IPV were type 1 30DU, type 2 32DU, type 3 45DU /0.5ml/per dose.

Inactivated Poliomyelitis Vaccine (Salk strains) was manufactured by Sanofi Pasteur D Ag contents /0.5ml/per dose were type 1 40DU, type 2 8DU, type 3 32DU.

This is a randomized, blind phase 3 clinical trial. Total 1200 infants (ages 60 days to 90 days) were selected, randomized to two groups (Sabin IPV and Salk IPV, each group n=600), infants in each group will be vaccinated with three doses of either Sabin IPV or Salk IPV respectively, one month apart.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age from 60 days to 90 days;
* Adults, parent(s) or guardians are able to understand and sign informed consent for participation;
* Participants or guardians are able to attend all planned clinical appointment and obey and follow all study instructions;
* Infants no vaccinated with poliovaccine or other preventive biologicals in recent 7 days;
* Axillary temperature ≤37℃.

Exclusion Criteria:

* Have medical record of participants or their family on allergy, convulsion, falling sickness, encephalopathy and psychopathy;
* Low platelet or bleeding disorder do not allow vaccination into the muscle;
* Have damaged or lower immunological function;
* Received blood, plasma or immunoglobulin treatment since birth;
* Have inborn abnormality, develop obstacles or clinical diagnostic serious chronic ( Down Syndrome, diabetes, sickle cell anemia or neural Guillain-Barre Syndrome );
* Have or be doubtful of following diseases: respiratory system diseases, acute infection or active chronic, cardiovascular diseases, liver and kidney diseases, skin diseases, HIV.

Exclusion Criteria for doses 2 and 3

* Have serious anaphylaxis or high fever, convulsion during first dose;
* Have any circus of Exclusion Criteria after Eligible for study;
* Have serious adverse event which related to previous vaccination; Withdrawal and Discontinuance Criteria;
* Received necessary or interference study drugs such as: immune-inhibition or immune-stimulating agents;
* Vaccinated with any other vaccine（except DTP）;
* Stop observation determined by investigator owing to occurring serious adverse event.

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The study on immunogenicity of Inactivated Poliomyelitis Vaccine made from Sabin Strains on Healthy infants | fours year
  Parallel study on comparison of sera protection rates (Neutralization antibody titer ≥1:8) of Sabin IPV and Salk IPV after three doses of vaccination.

SECONDARY OUTCOMES:
The study on efficacy of Inactivated Poliomyelitis Vaccine made from Sabin Strains on Healthy infants | One year
  Comparison of geometric mean titers (GMTs) of Sabin IPV and Salk IPV after three doses of vaccination
Mucosal Immunity - Comparison of intestinal excretion of polioviruses following one dose of tOPV after three doses of IPV | 30-60 days after third dose immunization
  One dose of tOPV was given after one month of third dose of IPV. The stool specimens were obtained at 0, 7, 14, 21, 28 days after OPV challenge. And determine the excretion rates of polioviruses.

CONTACTS AND LOCATIONS:
Overall Officials: Guoyang Liao, PH.D, Principal Investigator — Institute of Medical Biology, Chinese Academy of Medical Sciences; Yanping Li, MD, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control; Changgui Li, PHD, Principal Investigator — National Institute for the Control of Pharmaceutical and Biological Products, China
Locations (2):
- China (2):
  - Pingle Center for Disease Prevention and Control, Guilin, Guangxi
  - Bingyang Center for Disease Prevention and Control, Nanning, Guangxi

REFERENCES:
- [Derived] Ma L, Ying Z, Cai W, Wang J, Zhou J, Yang H, Gao J, Zhao Z, Liu J, Ouyang S, Song S, Shen F, Zhao R, Xu L, Dai X, Wu Y, Li W, Li C, Liao G. Immune persistence of an inactivated poliovirus vaccine derived from the Sabin strain: a 10-year follow-up of a phase 3 study. EClinicalMedicine. 2023 Sep 14;64:102151. doi: 10.1016/j.eclinm.2023.102151. eCollection 2023 Oct. PMID 37745024